CLINICAL TRIAL: NCT05343117
Title: Comparative Effectiveness of Palbociclib Based-therapy as Initial Endocrine Therapy Versus Palbociclib Based-therapy After Chemotherapy for HR+/HER2- Advanced Breast Cancer in Chinese Clinical Practice: a Real-world Study
Brief Title: Comparative Effectiveness of PAL Based-therapy as Initial ET Versus PAL Based-therapy After ChT for HR+/HER2- ABC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC3222
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Hormone Receptor Positive Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Palbociclib based-therapy as initial endocrine therapy: Adult patients with HR+/HER2- advanced breast cancer who received palbociclib based-therapy as initial endocrine therapy from August 1, 2018 to December 31, 2023.
  Interventions: Drug: Palbociclib based-therapy as initial endocrine therapy
- Palbociclib based-therapy after chemotherapy: Adult patients with HR+/HER2- advanced breast cancer who received palbociclib based-therapy after chemotherapy from August 1, 2018 to December 31, 2023.
  Interventions: Drug: Palbociclib based-therapy after chemotherapy

INTERVENTIONS:
Drug: Palbociclib based-therapy as initial endocrine therapy — Palbociclib + aromatase inhibitor/fulvestrant (initial endocrine therapy)
  Groups: Palbociclib based-therapy as initial endocrine therapy
Drug: Palbociclib based-therapy after chemotherapy — Palbociclib + aromatase inhibitor/fulvestrant (after chemotherapy)
  Groups: Palbociclib based-therapy after chemotherapy

SUMMARY:
A multi-center non-interventional observational study led by the Cancer Hospital Chinese Academy of Medical Sciences to compare the effectiveness of palbociclib based-therapy as initial endocrine therapy versus palbociclib based-therapy after chemotherapy for HR+/HER2- advanced breast cancer.

DETAILED DESCRIPTION:
This study is designed to be a multi-center non-interventional observational study led by the Cancer Hospital Chinese Academy of Medical Sciences. The target populations of this study are patients with HR+/HER2- advanced breast cancer who received palbociclib based-therapy as initial endocrine therapy or palbociclib based-therapy after chemotherapy from August 1, 2018 to December 31, 2023. It is expected to enroll 400 subjects in this study. The subjects' data such as demographics and other baseline characteristics, medications, prognosis, will be collected in a mixed manner, and statistical analysis of data will be conducted to compare the effectiveness outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, female (retrospective part);
2. Histologically or cytologically confirmed recurrent or metastatic HR+/HER2- breast cancer, if there was metastatic pathology, the histological pathology of metastases should prevail (retrospective part);
3. Received palbociclib in combination with endocrine therapy as initial therapy in the first line and received at least 1 cycle; or received systemic chemotherapy in the first line followed by sequential palbociclib in combination with endocrine therapy and received at least 1 cycle (retrospective part);
4. The follow-up time was not less than 3 months after the initiation of palbociclib in combination with endocrine therapy (retrospective part);
5. Age ≥ 18 years, female (prospective part);
6. Histologically or cytologically confirmed recurrent or metastatic HR+/HER2- breast cancer, if there is metastatic pathology, the histological pathology of metastases should prevail (prospective part);
7. ECOG PS ≤ 2, and expected survival of more than half a year and no life-threatening visceral metastasis (prospective part);
8. Measurable disease (prospective part);
9. No or up to 1 regimen of chemotherapy for advanced breast cancer (prospective part);
10. The patient has good compliance, and needs to receive the treatment with the palbociclib-based therapy according to the condition (prospective part);
11. Normal function of major organs and hematopoietic function, i.e. meeting the following criteria: Blood cell count criteria should be in accordance with: (no blood transfusion and blood products, no G-CSF and other hematopoietic stimulating factors for correction in recent 14 days): Hemoglobin (HB) ≥ 80 g/L; Neutrophils (ANC) ≥ 1.5 × 10^9/L; Platelet (PLT) ≥ 75 × 10^9/L. Liver function, renal function and electrolytes meeting the following criteria: Total bilirubin (TBIL) < 1.5 upper limit of normal (ULN), ≤ 3 ULN for patients with liver metastases; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 ULN, and ≤ 5 ULN for patients with liver metastases; Serum Cr ≤ 1.5 ULN or endogenous creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); Electrolytes: magnesium ≥ lower limit of normal (LLN) (prospective part);
12. The patient is compliant and voluntarily accepts the treatment, follow-up visit, laboratory examination and other study procedures according to the doctor's prescription (prospective part).

Exclusion Criteria:

1. ≥ 2 prior lines of chemotherapy for advanced breast cancer (retrospective part);
2. Treatment with other CDK4/6 inhibitors (abemaciclib or ribociclib) or endocrine therapy only (retrospective part);
3. Life-threatening visceral metastases, and lesions not evaluable for response (prospective part);
4. Neutrophils < 1.5 × 10^9/L; platelets < 100 × 10^9/L; not improved after medication (prospective part);
5. Total bilirubin ≥ 1.5 times the upper limit of normal, AST and ALT ≥ 2 times the upper limit of normal; serum Cr ≥ 1.5 times the upper limit of normal (prospective part);
6. Have central nervous system or meningeal invasion (prospective part);
7. Women who are pregnant, lactating, or planning to have children (prospective part);
8. Received ≥ 2 prior lines of chemotherapy for advanced breast cancer (prospective part);
9. Treatment with other CDK4/6 inhibitors (abemaciclib or ribociclib) or endocrine therapy only (prospective part);
10. Concomitant poorly controlled serious illness, major surgery, or history of other malignancy within 5 years (prospective part);
11. Other conditions that the investigator considers inappropriate for inclusion (prospective part).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with HR+/HER2- advanced breast cancer who received palbociclib based-therapy as initial endocrine therapy versus palbociclib based-therapy after chemotherapy from August 1, 2018 to December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  It is defined as the time (months) from the start of palbociclib based-therapy to progressive disease or all-cause mortality. The progressive disease is determined by clinicians based on the results of clinical evaluation, laboratory tests, imaging or pathological examinations. Patients who have not died or have not experienced progressive disease will be censored at the beginning of next-line treatment or at the last visit during the study period.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  ORR is defined as the proportion of patients with complete response (CR) or partial response (PR) reported by doctors among all patients with response data available.
Disease control rate (DCR) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  DCR is defined as the proportion of patients who have reached CR, PR, or stable disease (SD) reported by the doctors among all patients with response data available.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (9):
- China (9):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - The Third Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - The Fourth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - PLA Strategic Support Force Characteristic Medical Center, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei